CLINICAL TRIAL: NCT05557214
Title: Reducing Unnecessary Antibiotic Prescriptions in Primary Healthcare in Saskatchewan by Identifying High Prescribers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to execute data sharing agreement with Ministry of Health.
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Principal Investigator, Jason Vanstone, Research Scientist, Saskatchewan Health Authority - Regina Area
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB-22-38
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Upper Respiratory Tract Infections
Keywords: audit and feedback; antimicrobials; primary healthcare
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audit and Feedback Letter (Experimental): This group will receive 2 audit and feedback letters and a study closure letter.
  Interventions: Behavioral: Audit and Feedback Letter
- No Audit and Feedback Letter (No Intervention): This group will only receive a study closure letter.

INTERVENTIONS:
Behavioral: Audit and Feedback Letter — Physicians in the Audit and Feedback Letter Arm will receive an initial letter indicating their high prescriber status with guidance on reducing unnecessary antimicrobial use. They will also receive a follow-up letter at the 6 month mark indicating any change in prescribing habits. There will be a study closure letter mailed at the 12 month mark.
  Arms: Audit and Feedback Letter

SUMMARY:
Approximately 90% of antibiotics are prescribed in primary healthcare (PHC) in Canada (Public Health Agency of Canada, 2020), making this an important sector for antimicrobial stewardship. Upper respiratory tract infections (URTIs) represent a common indication in PHC for which antibiotics are often prescribed unnecessarily (Leis et al, 2020; Schwartz et al., 2020). Reducing unnecessary antibiotic treatment in this sector is a vital part of contributing to minimizing the global burden of antibiotic resistance.

The goal of this research project is to reduce the number of antibiotic prescriptions among family physicians identified as high prescribers in Saskatchewan. To achieve this, the investigators will send letters to the top 25th percentile of high prescribers in PHC. The letters will contain data indicating the prescribers high antimicrobial usage as well as guidance for reducing unnecessary prescriptions and promoting appropriate lengths of prescriptions for upper respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* must be a practicing family physician in Saskatchewan
* top 25th percentile of antimicrobial prescribers

Exclusion Criteria:

* fewer than 12 months of historical prescribing data available

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Total Antibiotic Prescriptions | 12 months
  Total number of antibiotic prescriptions compared to covariate-adjusted baseline number of prescriptions prior to the intervention.

SECONDARY OUTCOMES:
Total Prolonged-Duration Prescription | 12 months
  Number of prescriptions longer than 7 days.
Total Days of Therapy | 12 months
  Number of days of therapy of antimicrobials for each provider.
Antibiotic Cost | 12 months
  Total cost of prescribed antibiotics.
Total Specific Antibiotic Prescriptions | 12 months
  Number of prescriptions for specific antibiotics.

IPD SHARING:
Plan to Share IPD: No
Deidentified aggregate data will be shared via a published manuscript at the conclusion of the study.

REFERENCES:
- [Background] Leis JA, Born KB, Ostrow O, Moser A, Grill A. Prescriber-led practice changes that can bolster antimicrobial stewardship in community health care settings. Can Commun Dis Rep. 2020 Jan 2;46(1):1-5. doi: 10.14745/ccdr.v46i01a01. eCollection 2020 Jan 2. PMID 31930218
- [Background] Schwartz KL, Langford BJ, Daneman N, Chen B, Brown KA, McIsaac W, Tu K, Candido E, Johnstone J, Leung V, Hwee J, Silverman M, Wu JHC, Garber G. Unnecessary antibiotic prescribing in a Canadian primary care setting: a descriptive analysis using routinely collected electronic medical record data. CMAJ Open. 2020 May 7;8(2):E360-E369. doi: 10.9778/cmajo.20190175. Print 2020 Apr-Jun. PMID 32381687